CLINICAL TRIAL: NCT06566001
Title: Comparative Study Between Socket Shield Technique Versus Allograft Buccal Sheet Technique on Alveolar Bone Resorption After Immediate Implant Placement in Esthetic Region ( Randomised Clinic Trial)
Brief Title: Comparative Study Between Socket Shield Technique Versus Allograft Buccal Sheet Technique on Alveolar Bone Resorption After Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Hatem Rafaat, cairo, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422019476446
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2022-03

CONDITIONS: Bone Loss in Jaw
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group 11 patients (Experimental): socket shield technique 11 patients
  Interventions: Procedure: control group
- study group 11 patients (Experimental): allogenic buccal sheet technique 11 patients
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: control group — socket shield technique and allogenic bone graft

SUMMARY:
22 patient where divided randomly into 2 groups : control group did dental implant utilizing socket shield , while study group did dental implant with allogenic bone graft there is no significant bone loss between the two groups after 4 month follow up

ELIGIBILITY:
Inclusion Criteria:

- patient has remaining root in upper anterior without lesion

Exclusion Criteria:

periapical lesion under the tooth

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
measure bone loss by CBCT | 4 month
  Measure bone loss by CBCT mm

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt